CLINICAL TRIAL: NCT07073274
Title: EEG Analysis During Anesthesia for Day Case Gastroscopy and/or Colonoscopy
Brief Title: EEG During Gastroscopy and/or Colonoscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HUB2025185
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Endoscopy of Stomach (Procedure); Colonoscopy (Procedure); Continuous Processed Electroencephalogram (Procedure)
Keywords: Anesthesia; EEG; Burst suppression; gastroscopy; colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EEG monitoring (Other): Continuous EEG monitoring
  Interventions: Diagnostic Test: EEG analysis

INTERVENTIONS:
Diagnostic Test: EEG analysis — All patients will have a continous recording of their EEG during anesthesia

SUMMARY:
During anesthesia, EEG shows specific and significant changes according to the depth of anesthesia and the drugs used. Endoscopic procedures like gastroscopies or colonoscopies are usually done on an outpatient basis using essentially propofol for sedation or anesthesia. Preliminary reports have shown that the depth of anesthesia during these procedures may be very deep resulting even in a burst suppression pattern on the EEG.

In this study, frontal EEG will be recorded continuously using a Root - Sedline device (Masimo, US). Anesthesiologists will be free to use the medications and dosage they judge appropriate. The attending anesthesiologist will be blinded to the EEG. Medications and dosages will be recorded, as well as processed EEG data from the Sedline and the raw EEG. Primary outcome is the % of time spend in specific range of patient state index (PSI 0-10; 10-20; 20-30; 30-40; 40-50; 5-60; 60-70; 70-80; 80-90; 90-100) as well as the % of time spent in burst suppression.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing gastroscopy and or colonoscopy in a outpatient setting under sedation or general anesthesia

Exclusion Criteria:

* Patients < 18 years
* altered renal function, Glomerular filtration rate < 50 mL/min/m2
* altered hepatic tests, > 1.5 * upper normal limit
* Any form of hepatic cirrhosis
* Presence of oesophageal varices
* Any neurological pathology rendering EEG analysis non reliable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Burst suppression | 90 min
  Percentage of time spent in burst suppression
PSI | 90 min
  Percentage of time spent in each PSI range

CONTACTS AND LOCATIONS:
Locations (1):
- H.U.B _ Hôpital Erasme, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] John ER, Prichep LS, Kox W, Valdes-Sosa P, Bosch-Bayard J, Aubert E, Tom M, di Michele F, Gugino LD. Invariant reversible QEEG effects of anesthetics. Conscious Cogn. 2001 Jun;10(2):165-83. doi: 10.1006/ccog.2001.0507. PMID 11414713